CLINICAL TRIAL: NCT07169136
Title: Effects of Glucagon-like Peptide-1 (GLP-1) Agonist in Neuro-reproductive Function in Obese Adolescent Females With Polycystic Ovary Syndrome (PCOS)
Status: Recruiting | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Camila Pereira-Eshraghi, MD., Nemours Children's Clinic
Other Study IDs: 25-014
Record Dates: First submitted 2025-08-19; First posted 2025-09-11 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Polycystic Ovarian Syndrome in Adolescent Females; Obesity (Disorder)
Keywords: PCOS; Obesity; Adolescent Female; irregular menstrual cycles
MeSH Terms: conditions — Obesity; Menstruation Disturbances | interventions — Glucagon-Like Peptide-1 Receptor Agonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Females ages 12 to 18 years, at least 2 years post-menarche, with obesity and PCOS..: Females ages 12 to 18 years, at least 2 years post-menarche, with obesity (BMI equal to or more than the 95th percentile for age) and with PCOS, by NIH criteria: oligomenorrhea (menstrual cycles <21 or >35 days) [4] and hyperandrogenism (testosterone level or free androgen index (FAI) > refence range for tanner stage) and in good overall health. FAI is calculated as total testosterone*100/sex hormone binding globulin.
  Interventions: Drug: GLP-1 Receptor Agonists

INTERVENTIONS:
Drug: GLP-1 Receptor Agonists — Weekly subcutaneous Semaglutide.

SUMMARY:
The prevalence of childhood obesity in the United States has more than tripled in the past four decades affecting one in every five adolescent girls and is disproportionally higher among racial and/or ethnic minorities. Normal puberty onset and progression is dependent on normal hypothalamic-pituitary-gonadal (HPG) axis which is affected by whole body metabolism. Gonadotropin-releasing hormone (GnRH) and gonadotropins, LH and FSH, are released in a pulsatile manner for appropriate sex steroids production and gonadal function. Proper pulsatility in the GnRH system is disrupted by a significant change in energy balance such as in obesity. Polycystic Ovary Syndrome (PCOS) is the most common neuroendocrine dysfunction in women of reproductive age. Glucagon-like peptide-1 (GL-1), a peptide hormone secreted by the intestinal enteroendocrine L-cells following glucose and fat intake, stimulates insulin release by the pancreas in response to glucose, decreases gastric emptying and inhibits glucagon secretion. GLP-1 receptors are present in the hypothalamic nuclei and pituitary gland; and it is thought that GLP-1 may directly stimulate GnRH secretion and partially regulate reproduction. In animal studies, GLP-1 was found to stimulate GnRH secretion, to regulate kisspeptin (Kiss-1) mRNA and GnRH mRAN expression. GLP-1 receptor agonists are FDA-approved to treat adults and adolescents with obesity. Although the impact of GLP-1 receptor agonists in reproductive health has been investigated in preclinical trials, and in men with obesity and functional hypogonadism, no studies to date have investigated the impact of GLP-1 receptor agonists in female neuroendocrine function, particularly in youth. The goal of this proposal is to gather critical preliminary data to investigate, in a group of obese adolescent females with PCOS, the impact of GLP-1 agonist administration in addition to lifestyle modifications on the neuroendocrine rhythms - LH frequency and amplitude (principal); body composition, adiposity; and carbohydrate metabolism and insulin sensitivity. To accomplish these aims, we will recruit a cohort of up to 20 adolescents ages 12-18 years, at least 2 years post-menarche, with obesity, PCOS, by NIH criteria, without carbohydrate intolerance and in otherwise good health. Research volunteers will be advised on lifestyle modifications of diet and exercise as per routine, and a GLP-1 agonist will be started according to the product's label as per FDA guidelines in children with obesity. Medication will be titrated to maximal therapeutic dose, as per routine clinical practice. Participants will be treated for a total of 16 weeks. Neuroendocrine rhythms pre- and post-treatment will be compared.

DETAILED DESCRIPTION:
The prevalence of childhood obesity in the United States has more than tripled in the past four decades affecting one in every five adolescent girls and is disproportionally higher among racial and/or ethnic minorities. Normal puberty onset and progression is dependent on normal hypothalamic-pituitary-gonadal (HPG) axis which is affected by whole body metabolism. Gonadotropin-releasing hormone (GnRH) and gonadotropins, LH and FSH, are released in a pulsatile manner for appropriate sex steroids production and gonadal function. Proper pulsatility in the GnRH system is disrupted by a significant change in energy balance such as in obesity. Polycystic Ovary Syndrome (PCOS) is the most common neuroendocrine dysfunction in women of reproductive age.

Glucagon-like peptide-1 (GL-1), a peptide hormone secreted by the intestinal enteroendocrine L-cells following glucose and fat intake, stimulates insulin release by the pancreas in response to glucose, decreases gastric emptying and inhibits glucagon secretion. GLP-1 receptors are present in the hypothalamic nuclei and pituitary gland; and it is thought that GLP-1 may directly stimulate GnRH secretion and partially regulate reproduction. In animal studies, GLP-1 was found to stimulate GnRH secretion, to regulate kisspeptin (Kiss-1) mRNA and GnRH mRAN expression. GLP-1 receptor agonists are established diabetes drugs that are also promising anti-obesity drugs and are FDA-approved to treat adults and adolescents with obesity. Although the impact of GLP-1 receptor agonists in reproductive health has been investigated in preclinical trials, and in men with obesity and functional hypogonadism, no studies to date have investigated the impact of GLP-1 receptor agonists in female neuroendocrine function, particularly in youth.

The goal of this proposal is to gather critical preliminary data to investigate, in a group of obese adolescent females with oligomenorrhea due to PCOS, the impact of GLP-1 agonist administration in addition to lifestyle modifications on -

Aim 1. neuroendocrine rhythms - LH frequency and amplitude (principal); Aim 2. body composition; Aim 3. carbohydrate metabolism and insulin sensitivity. The investigators hypothesize that 16 weeks intervention with a GLP-1 agonist will result in improvement of gonadotropin release patterns.

To accomplish these aims, the investigators will recruit a cohort of up to 20 adolescents ages 12-18 years, at least 2 years post-menarche, with obesity (BMI-for-age equal to or more than the 95th percentile), with PCOS, by NIH criteria: oligomenorrhea and hyperandrogenism (testosterone level or free androgen index > refence range for tanner stage.), without carbohydrate intolerance and in otherwise good health. Research volunteers will be advised on lifestyle modifications of diet and exercise as per routine, and a GLP-1 agonist will be started according to the product's label as per FDA guidelines in children with obesity. Medication will be titrated to maximal therapeutic dose, as per routine clinical practice, and continued for a total of 16 weeks.

Principal Study Outcomes

1. Reproductive measures will include change in: LH pulse frequency and amplitude, average levels of LH and FSH, and estradiol, total testosterone
2. Body composition will be measured by dual x-ray absorptiometry (DXA) scan
3. Carbohydrate metabolism and insulin sensitivity will be measured by HOMA-IR (using fasting insulin and glucose levels).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PCOS, by NIH criteria: oligomenorrhea (menstrual cycles <21 or >35 days) and hyperandrogenism (testosterone level or free androgen index (FAI) > refence range for tanner stage) and in good overall health
* Obesity (equal to or more than the 95th percentile)
* Females ages 12 to 18 years, at least 2 years post-menarche
* Participants has persistent symptoms of PCOS and obesity despite lifestyle modifications for at least 4 months.

Exclusion Criteria:

* Has abnormal thyroid function tests at Screening.
* Has suspected or known Diabetes mellitus, impaired fasting glucose, or elevated hemoglobin A1c.
* Has non-classic congenital adrenal hyperplasia.
* Has hyperprolactinemia.
* Has a known history or family history of medullary thyroid carcinoma or MEN2 and history of pancreatitis
* Participants receiving prior treatment with metformin, GLP-1 agonists, oral contraception pills, progesterone, or other insulin sensitizers for at least 6 weeks prior to Screening.
* Is currently pregnant or has been pregnant.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescent females with Obesity and PCOS.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in LH pulse frequency after 4 months of GLP-1 agonist use. | Blood sampling will occur at study enrollment and then 4 months post intervention.
  LH will be obtained every 20 minutes overnight. LH will be measured using a chemiluminescence assay. Pulse frequency will be calculated using mathematical deconvolution analysis.
Change in average levels of LH and FSH after 4 months of GLP-1 agonist use. | Blood sampling will occur at study enrollment and then 4 months post intervention.
  LH and FSH will be measured using a chemiluminescence assay.
Change in average levels of Total testosterone and Estradiol after 4 months of GLP-1 agonist use. | Blood sampling will occur at study enrollment and then 4 months post intervention.
  Total testosterone and estradiol will be measured by liquid chromatography-mass spectrometry
Change in average levels of progesterone after 4 months of GLP-1 agonist use. | Blood sampling will occur at study enrollment and then 4 months post intervention.
  Progesterone will be measured using immunoassay.
Change in LH amplitude. | Blood sampling will occur at study enrollment and then 4 months post intervention.
  LH will be obtained every 20 minutes overnight. LH will be measured using a chemiluminescence assay. Pulse amplitude will be calculated using mathematical deconvolution analysis.

SECONDARY OUTCOMES:
Body composition will be measured by dual x-ray absorptiometry (DXA) scan. | At enrollment and 4 months post intervention.
  Body composition will be measured by DEXA (Hologic Discovery A)
Carbohydrate metabolism and insulin sensitivity will be analyzed. | Sampling will occur at enrollement and 4 months post intervention.
  Carbohydrate metabolism and insulin sensitivity will be measured by HOMA-IR (using fasting insulin and glucose levels).

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD captured during the study trial will be shared deidentified.

REFERENCES:
- [Background] McCartney CR, Campbell RE. Abnormal GnRH Pulsatility in Polycystic Ovary Syndrome: Recent Insights. Curr Opin Endocr Metab Res. 2020 Jun;12:78-84. doi: 10.1016/j.coemr.2020.04.005. Epub 2020 Apr 23. PMID 32676541
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Ruffing KM, Koltun KJ, De Souza MJ, Williams NI. Moderate Weight Loss is associated with Reductions in LH Pulse Frequency and Increases in 24-hour Cortisol with no change in Perceived Stress in Young Ovulatory Women. Physiol Behav. 2022 Oct 1;254:113885. doi: 10.1016/j.physbeh.2022.113885. Epub 2022 Jun 16. PMID 35718216
- [Background] McCartney CR, Prendergast KA, Blank SK, Helm KD, Chhabra S, Marshall JC. Maturation of luteinizing hormone (gonadotropin-releasing hormone) secretion across puberty: evidence for altered regulation in obese peripubertal girls. J Clin Endocrinol Metab. 2009 Jan;94(1):56-66. doi: 10.1210/jc.2008-1252. Epub 2008 Oct 28. PMID 18957503